CLINICAL TRIAL: NCT05195476
Title: Neural Correlates of Compulsivity
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: International OCD Foundation (Unknown)
Responsible Party: Principal Investigator, Amy Rapp, Assistant Professor of Clinical Medical Psychology (in Psychiatry), Columbia University
Other Study IDs: 7867
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Compulsivity; Obsessive-Compulsive Disorder; Exposure and Response Prevention; Electroencephalogram
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals diagnosed with OCD: Individuals diagnosed with OCD
- Healthy controls: Individuals who have not been diagnosed with any psychiatric disorders

SUMMARY:
This study aims to collect data from individuals with obsessive-compulsive disorder (OCD) and healthy controls in order to clarify how learning strategies are employed differently by individuals with compulsive psychopathology and healthy individuals. Behavioral and electroencephalogram (EEG) data will be collected during one experimental reinforcement learning tasks from participants diagnosed with OCD (n = 30) and healthy controls (n = 30). Computational modeling, an advanced data analytic approach that can directly link neural measures with behavior, will be used to quantify learning processes. These parameters then will be related to measures of neural events obtained using EEG, a neuroimaging method that has high temporal resolution, to test for evidence of neurocognitive alterations.

DETAILED DESCRIPTION:
Learning and decisions making are thought to be directed by multiple parallel cognitive systems. These systems account for automatic, inflexible responding to stimuli, as well as more deliberate, effortful representations of relationships in an environment. It has long been suggested than an imbalance in these cognitive control systems explains the emergence of compulsivity, a trait in which behaviors persist despite adverse outcomes. Compulsivity is a characteristic of a number of psychological disorders, however, current theories of how abnormalities in cognitive systems involved in learning and decision making lead to the onset of these disorders remain incomplete.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-50 years of age
* English-speaking
* Capacity to provide informed consent
* Primary diagnosis of OCD with at least moderate severity

Exclusion Criteria:

* Current or lifetime history of psychiatric disorders other than OCD that may increase the risk of participation
* History of any significant medical condition that may increase the risk of participation
* Alcohol or substance use disorder in the past year
* Exposure and response prevention for OCD within the last six weeks
* Currently taking psychotropic medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals diagnosed with OCD and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Neural Activity | One-time study visit
  EEG will be recorded while participants complete computerized reinforcement learning tasks at one study visit

CONTACTS AND LOCATIONS:
Overall Officials: Amy Rapp, PhD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States